CLINICAL TRIAL: NCT05387954
Title: Transcatheter Patent Foramen Ovale (PFO) Closure, Oral Anticoagulants or Antiplatelet Therapy After PFO-associated Stroke in Patients Between 60 and 80 Years Old : a Randomised Controlled Trial.
Brief Title: PFO Closure, Oral Anticoagulants or Antiplatelet Therapy After PFO-associated Stroke in Patients Aged 60 to 80 Years
Acronym: CLOSE-2
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Ministry of Health, France (Other Government); W.L.Gore & Associates (Industry); Abbott (Industry); Occlutech International AB (Industry); Centre Hospitalier St Anne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: APHP211041; 2021-A03197-34 (Other: IDRCB); PHRC-20-0680 (Other: Ministry of health (France))
Record Dates: First submitted 2022-05-04; First posted 2022-05-24 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Cryptogenic Ischemic Stroke; Patent Foramen Ovale
Keywords: Ischemic stroke; Cryptogenic stroke; Patent foramen ovale; Atrial septal aneurysm; Transcatheter PFO closure; Oral anticoagulants; Antiplatelet therapy; Randomized clinical tria
MeSH Terms: conditions — Ischemic Stroke; Foramen Ovale, Patent | interventions — Factor Xa Inhibitors

STUDY DESIGN:
Intervention Model Description: PFO closure + antiplatelet therapy versus antiplatelet therapy alone Oral anticoagulants versus antiplatelet therapy
Who Masked: Outcomes Assessor
Masking Description: The clinical event adjudication committee will blind to the treatment allocated by randomization.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Antiplatelet therapy (Active Comparator): Aspirin OR clopidogrel
  Interventions: Drug: Antiplatelet therapy
- Oral anticoagulants, Direct-Acting (Experimental): Apixaban (5mg twice a day) OR Dabigatran (150 mg twice a day) OR Rivaroxaban (20 mg once a day)
  Interventions: Drug: Oral Anticoagulant, Direct-Acting
- PFO closure (Experimental): PFO closure followed by dual antiplatelet therapy (aspirin 75 mg/d + clopidogrel 75 mg/d) for 3 months, then by single antiplatelet therapy by aspirin or clopidogrel
  Interventions: Procedure: Transcatheter PFO closure; Drug: Antiplatelet therapy

INTERVENTIONS:
Procedure: Transcatheter PFO closure — PFO closure followed by dual antiplatelet therapy (aspirin 75 mg/d + clopidogrel 75 mg/d) for 3 months, then by single antiplatelet therapy by aspirin or clopidogrel until the end of the study.
  Other Names: •Each device for PFO closure must have the CE mark; •and be approved by the Interventional Cardiology Committee
  Arms: PFO closure
Drug: Oral Anticoagulant, Direct-Acting — Apixaban (5mg twice a day) OR Dabigatran (150 mg twice a day) OR Rivaroxaban (20 mg once a day)
  Arms: Oral anticoagulants, Direct-Acting
Drug: Antiplatelet therapy — Patients randomized to this arm will receive antiplatelet therapy throughout the study : aspirin 75 mg/d + clopidogrel 75 mg/d) for 3 months, then single antiplatelet therapy by aspirin or clopidogrel
  Arms: Antiplatelet therapy; PFO closure

SUMMARY:
To assess whether PFO closure plus antiplatelet therapy is superior to antiplatelet therapy alone and whether oral anticoagulant therapy is superior to antiplatelet therapy to prevent stroke recurrence in patients aged 60 to 80 years with a PFO with large shunt (> 20 microbubbles) or a PFO associated with an ASA (> 10 mm), and an otherwise unexplained ischemic stroke.

DETAILED DESCRIPTION:
The CLOSE trial (NCT00562289, NEJM 2017) has unambiguously demonstrated the superiority of patent foramen ovale (PFO) closure over antiplatelet therapy alone in patients aged up to 60 years with a PFO associated with an atrial septal aneurysm (ASA) or a large right-to-left shunt (so-called "high-risk PFO"), and an otherwise unexplained ischemic stroke. Oral anticoagulant therapy is also a logical approach assuming that PFO-related strokes are due to paradoxical embolism which implies a venous source of embolism, or to direct embolization of a thrombus formed at the atrial level. The CLOSE trial also suggested that oral anticoagulants might reduce stroke recurrence compared to aspirin.

There is accumulating evidence that presence of a PFO is significantly associated with cryptogenic stroke in patients over 60 years. Cryptogenic ischemic strokes represent about one third of all ischemic strokes in patients older than 60 years. However, the optimal therapeutic strategy in patients older than 60 years with a PFO and an otherwise unexplained ischemic stroke is unknown, because these patients were excluded from randomized trials.

The hypothesis tested in this trial is that transcatheter PFO closure plus long-term antiplatelet therapy is superior to antiplatelet therapy alone and that oral anticoagulant therapy is superior to antiplatelet therapy to prevent recurrent stroke in patients aged 60 to 80 years who have a high-risk PFO and a recent otherwise unexplained ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman aged 60 to 80 years.
* Recent (≤ 6 months) ischemic stroke confirmed by cerebral imaging regardless of symptom duration.
* Absence of a more probable cause of stroke than PFO after a standardized etiological work-up (see addenda).
* Presence of a PFO with at least 1 of the 2 following characteristics:

  * PFO with large shunt > 20 microbubbles appearing in the left atrium during at least one of the 3 cardiac cycles after opacification of the right atrium, detected spontaneously or during provocative manoeuvers, on contrast transthoracic (TTE) or transoesophageal (TOE) echocardiography. The diagnosis of PFO by contrast TEE must be confirmed by contrast TOE showing a right-to-left passage of the contrast material across the PFO.
  * PFO with ASA on transoesophageal echocardiography: excursion >10 mm
* Affiliation to a French Health Insurance system. Informed consent.

Exclusion Criteria:

* Life expectancy < 4 years.
* Contraindication to both experimental treatments (PFO closure, oral anticoagulant therapy) or to the reference treatment (antiplatelet therapy) (see paragraph 20.5).
* Indication to long-term anticoagulant therapy.
* mRS >= 3.
* Presence of other medical conditions that would lead to inability to complete the study or interfere with the assessment of outcomes.
* Previous surgical or transcatheter treatment of PFO or ASA. Expected impossible follow-up or poor compliance.
* Patient unable to understand the informed consent form. Patient under tutorship, curatorship, or legal protection.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 792 (Estimated)
Dates: Start 2023-07-07 (Actual); Primary Completion 2031-07-07 (Estimated); Study Completion 2031-07-07 (Estimated)

PRIMARY OUTCOMES:
Time to recurrent stroke (ischemic or hemorrhagic fatal or non-fatal) | From date of randomization until the date of first recurrent stroke, assessed from up to 4 years (for the last patient included) to up to 8 years (for the first patient included)
  Stroke: sudden onset of focal neurological symptoms related to a disturbance of the cerebral circulation.
  Ischemic stroke : at least one of the following criteria:
  * Sudden onset of focal neurological symptoms with the presence of cerebral infarction in the appropriate territory on brain imaging (CT or MRI), regardless of the duration of symptoms (less than or more than 24 hours).
  * Sudden onset of focal neurological symptoms lasting more than 24 hours, with no apparent cause other than cerebral ischemia.
  Intracerebral hemorrhage: sudden onset of focal neurological symptoms with the presence of cerebral hemorrhage in the appropriate territory on brain imaging (CT or MRI), regardless of the duration of symptoms (less than or more than 24 hours) and regardless of the cause of the hemorrhage (spontaneous or secondary to trauma, tumour or another cause).
  Unknown type of stroke : the type of stroke cannot be determined with certainty and the symptoms last more than 24 hours.

SECONDARY OUTCOMES:
Time to disabling stroke | From date of randomization until the date of first recurrent disabling stroke, assessed from up to 4 years (for the last patient included) to up to 8 years (for the first patient included)
  mRS score greater than or equal to 3, with an increase of at least 2 points compared to the last mRS score before the stroke.
Time to ischemic stroke | From date of randomization until the date of first recurrent ischemic stroke, assessed from up to 4 years (for the last patient included) to up to 8 years (for the first patient included)
  At least one of the following criteria:
  * Sudden onset of focal neurological symptoms with the presence of cerebral infarction in the appropriate territory on brain imaging (CT or MRI), regardless of the duration of symptoms (less than or more than 24 hours).
  * Sudden onset of focal neurological symptoms lasting more than 24 hours, with no apparent cause other than cerebral ischemia.
Time to ischemic stroke or systemic embolism | From date of randomization until the date of first recurrent ischemic stroke or systemic embolism, assessed from up to 4 years (for the last patient included) to up to 8 years (for the first patient included)
  Clinical features related to embolism usually affecting a limb, mesenteric, splenic, or renal artery. The diagnosis of embolism must be confirmed by appropriate investigations.
Time to transient ischemic attack, | From date of randomization until the date of first transient ischemic attack, assessed from up to 4 years (for the last patient included) to up to 8 years (for the first patient included)
  Sudden onset of neurological symptoms, presumed to be ischemic, resolving in less than 24 hours, clearly attributable to focal involvement of the central nervous system (or of the eye) with no signs of a corresponding recent cerebral infarction on brain imaging. The diagnosis of TIA will be confirmed by a neurologist, considering clinical data and brain imaging (MRI with diffusion sequence is recommended).
Time to vascular death | From date of randomization until the date of vascular death, assessed from up to 4 years (for the last patient included) to up to 8 years (for the first patient included)
  * death related to a cardiac or vascular cause.
  * death due to hemorrhage.
  * death due to pulmonary embolism.
  * sudden death: death occurring in less than 24 hours, unexpectedly in a subject in apparent good health and whose condition was stable or was improving.
  * death with no documented non-vascular cause.
  * fatal stroke: death occurring within 30 days of a stroke (ischemic or hemorrhagic).
Time to all-cause mortality | From date of randomization until the date of death, assessed from up to 4 years (for the last patient included) to up to 8 years (for the first patient included)
  Vascular (see definition) or nonvascular death: death due to a documented non-vascular cause (infection, cancer, accident, suicide, etc.).
Quality of life score | Every 6 months after randomization or up to 4 years (for the last patient included) to up to 8 years (for the first patient included)]
  Measured by using the European Quality Of Life (EQ-5D) auto-questionnaire. The digits for the five dimensions are combined into a 5-digit number that describes the patient's health state. The visual analogue scale (VAS) records the patient's self-rated health on a vertical axis from 0 (worst health) to 100 (best health)
Time to fatal, life-threatening or major hemorrhage, including intracerebral and Intracranial hemorrhage | From date of randomization until the date of first fatal,life-threatening or major hemorrhage,including intracerebral and Intracranial hemorrhage,assessed from up to 4 years(for the last patient included) to up to 8 years(for the first patient included)
  Life-threatening
  * Fatal hemorrhage.
  * Drop in hemoglobin by ≥ 5 g/dL (or drop in hematocrit by 15% or more in absolute value)
  * Symptomatic intracranial hemorrhage (confirmed by appropriate investigations, classified as cerebral hemorrhage, subarachnoid hemorrhage and subdural hematoma).
  * Transfusion ≥ 4 units of packed cells (or equivalent of whole blood)*.
  Major
  * Transfusion ≤ 3 units of packed cells (or equivalent of whole blood)*.
  * Requiring hospitalization (or prolonging hospitalization).
  * Requiring surgical treatment.
  * Intraocular hemorrhage with significant loss of vision.
  * Other hemorrhage responsible for significant disability according to the investigator.
Proportion of success of device implantation, of the procedure and of PFO closure, | 6 months after PFO closure
  * Success of device implantation: deployment of the device in the appropriate place and removal of the placement system.
  * Success of the procedure: successful implantation with no complications before the patient's discharge.
  * Success of PFO closure: success of the procedure with no residual shunt or minimal residual shunt on echocardiography performed 6 months after the procedure.
Time to ischemic stroke recurrence according to the presence of a residual shunt | From date of PFO closure until the date of first ischemic stroke recurrence, assessed from up to 4 years (for the last patient included) to up to 8 years (for the first patient included), according to the presence of residual shunt]
  From control echocardiography after PFO closure to the end of the patient's follow-up
Time to new-onset atrial fibrillation | From date of randomization until the date of new-onset atrial fibrillation, assessed from up to 4 years (for the last patient included) to up to 8 years (for the first patient included)]
  Atrial fibrillation lasting at least 30 seconds
Proportion of fatal, life-threatening or major procedure- or device-related complications | Within 4 weeks following the procedure (PFO closure)
  Life-threatening
  * Cardiac perforation with tamponade requiring emergency drainage.
  * Cerebral air embolism responsible for acute neurological disorders
  * Embolization of the device.
  * Life-threatening hematoma at the puncture site or retroperitoneal.
  * Complications of general anesthesia or TOE requiring intensive care and/or surgical operation.
  Major
  * Hemorrhage at the puncture site or retroperitoneal requiring transfusion or surgery.
  * Arteriovenous fistula, pseudoaneurysm requiring surgery.
  * Peripheral nerve lesion with disabling neurological deficit persisting > 1 month.
  * Cardiac arrhythmias (particularly AF) during catheterization or post-procedure requiring treatment >= 1 month.
  * Infective endocarditis.
  * Asymptomatic late thrombosis of the device.
  * Any device-related complication requiring surgery.
  * Any other complication related to the transcatheter treatment or anesthesia, considered to be major by the investigator.
Costs | Within 48 months after randomization
  Costs will be estimated from the viewpoint of the healthcare system (hospital admission, transportation, study interventions, emergency room visit without admission,consultations,imaging)
Incremental cost-utility ratio at 4 years (ICUR) | Within 48 months after randomization
  The incremental cost-utility ratio (ICUR) will be calculated as difference in costs (between groups)/difference in QALYs (Quality-Adjusted Life Year) between groups.
  The QALYs will be constructed with the EuroQoL-5D (EQ-5D) questionnaire and value sets

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Louis Mas, MD, Principal Investigator — GHU Psychiatrie et Neurosciences Paris; Gilles Chatellier, MD, Study Director — Hôpital Européen Georges-Pompidou
Locations (41):
- France (41):
  - CHU Amiens, Amiens
  - CH Arras, Arras
  - CHU Jean Minjoz, Besançon
  - CHU Bordeaux - GH Pellegrin, Bordeaux
  - CHRU La Cavale Blanche, Brest
  - HCL-Groupement Hospitalier Lyon Est, Bron
  - CHU Côte de Nacre, Caen
  - CHU Clermont Ferrand, Clermont-Ferrand
  - CH Sud Francilien, Corbeil-Essonnes
  - Hôpital Henri Mondor, Créteil
  - CHU Dijon-Hôpital François Mitterrand, Dijon
  - CH Grenoble-Site Nord, Grenoble
  - GPE Hospitalier La Rochelle-Ré-Aunis, La Rochelle
  - CH Versailles-Hôpital Mignot, Le Chesnay
  - CHU Bicêtre, Le Kremlin-Bicêtre
  - CHRU Lille-Hôpital Salengro, Lille
  - Hôpital de la Timone, Marseille
  - Grand Hôpital de l'Est Francilien, Meaux
  - Hôpital Gui de Chauliac, Montpellier
  - CHRU Nancy-Hôpital central, Nancy
  - CHU de Nice-Hôpital Pasteur, Nice
  - CHU Carémeau, Nîmes
  - CH Orsay, Orsay
  - APHP Hôpital Lariboisière, Paris
  - Hôpital Pitié Salpêtrière, Paris
  - GHU Paris Psychiatrie et Neurosciences, Paris
  - Groupe Hospitalier Paris Saint-Joseph, Paris
  - APHP Hôpital Bichat, Paris
  - Fondation Adolphe de Rothschild, Paris
  - CH Perpignan, Perpignan
  - CHU La Milétrie, Poitiers
  - Hôpital Novo, Pontoise
  - CHU Rennes-Hôpital Pontchaillou, Rennes
  - CHU Rouen-Hôpital Charles-Nicolle, Rouen
  - CH Yves Le Foll, Saint-Brieuc
  - CHU Nantes-Hôpital Nord Laennec, Saint-Herblain
  - CHU Saint-Etienne-Hôpital Nord, Saint-Priest-en-Jarez
  - Hôpital Hautepierre, Strasbourg
  - Hôpital Foch, Suresnes
  - CHU Toulouse-Hôpital Pierre Paul Riquet, Toulouse
  - CHRU Tours- Hôpital Bretonneau, Tours

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie results in publication could be shared. IPD detailed in the protocol of a planned metaanalysis could be shared
Supporting Information: Study Protocol, ICF
Time Frame: Two years after the last publication
Access Criteria: Data sharing must be accepted by the sponsor and the PI based on a scientific project and scientific involvement of the PI team. Collaboration will be fostered.
  Data sharing must respect the agreements made with funders.
  Teams wishing obtain IPD must meet the sponsor and PI team to present scientific (and commercial) purpose, IPD needed, format of data transmission, and timeframe. Technical feasability and financial support will be discussed before mandatory contractual agreement.
  Processing of shared data must comply with European General Data Protection Regulation (GDPR).